CLINICAL TRIAL: NCT04856930
Title: A Phase 2, Randomized, Double-Blind, Placebo Controlled Study to Evaluate the Efficacy and Safety of Imsidolimab (ANB019) in the Treatment of Subjects With Hidradenitis Suppurativa
Brief Title: A Study to Evaluate the Efficacy and Safety of Imsidolimab (ANB019) in the Treatment of Participants With Hidradenitis Suppurativa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANB019-208; 2021-001440-99 (EudraCT Number)
Record Dates: First submitted 2021-04-20; First posted 2021-04-23 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-04

CONDITIONS: Hidradenitis Suppurativa
Keywords: IL-36 receptor; Interleukin 36; Imsidolimab
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Imsidolimab 400/200 milligrams (mg) (Experimental): 400 milligrams (mg) of imsidolimab on Day 1 followed by 200 mg imsidolimab every 4 weeks by subcutaneous (SC) injection up to 48 weeks
  Interventions: Biological: Imsidolimab
- Imsidolimab 200/100 mg (Experimental): 400 milligrams (mg) of imsidolimab on Day 1 followed by 200 mg imsidolimab every 4 weeks by subcutaneous (SC) injection up to 48 weeks
  Interventions: Biological: Imsidolimab
- Placebo (Placebo Comparator): Placebo-controlled period: Participants received imsidolimab matching placebo on Day 1 and thereafter, every 4 weeks (Days 29, 57 and 85) by SC injection. The placebo-controlled period ended at Day 113 (Week 16).
  Extension period: Participants received imsidolimab at the same dose as placebo-controlled period, SC every 4 weeks (Days 113, 141, 169, and 197).
  After discontinuation from treatment, participants remained in the study for safety follow-up period of 8 weeks.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Imsidolimab — Humanized Monoclonal Antibody
  Other Names: ANB019
  Arms: Imsidolimab 200/100 mg; Imsidolimab 400/200 milligrams (mg)
Biological: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Efficacy and safety of imsidolimab (ANB019) in participants with Hidradenitis Suppurativa

DETAILED DESCRIPTION:
This is a Phase 2, multicenter, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of imsidolimab in adult participants with hidradenitis suppurativa (HS). This study will also characterize the pharmacokinetic (PK) profile of imsidolimab and explore the immune response to imsidolimab in participants with HS.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically confirmed diagnosis of active HS with a disease duration of greater than or equal to (≥) 6 months before Day 1.
2. HS lesions present in at least 2 distinct anatomical areas.
3. Total Abscess and inflammatory nodule (AN) count ≥ 5.
4. Draining fistulas less than or equal to (≤) 20.
5. Stable HS for at least 6 weeks prior to Day 1 visit.

Exclusion Criteria:

1. Concomitant dermatological or medical conditions that may interfere with the Investigators' ability to evaluate the participant's response to therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-12-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (34):
- United States (17):
  - Site 10-108, Birmingham, Alabama
  - Site 10-104, Fountain Valley, California
  - Site 10-119, Northridge, California
  - Site 10-102, Sacramento, California
  - Site 10-109, Coral Gables, Florida
  - Site 10-107, Largo, Florida
  - Site 10-111, Tampa, Florida
  - Site 10-110, Sandy Springs, Georgia
  - Site 10-101, Fort Gratiot, Michigan
  - Site 10-103, Portsmouth, New Hampshire
  - Site 10-115, Warwick, Rhode Island
  - Site 10-113, Greenville, South Carolina
  - Site 10-118, Houston, Texas
  - Site 10-112, Pflugerville, Texas
  - Site 10-117, San Antonio, Texas
  - Site 10-105, Norfolk, Virginia
  - Site 10-106, Spokane, Washington
- Canada (5):
  - Site 11-106, Calgary, Alberta
  - Site 11-103, Cobourg, Ontario
  - Site 11-102, Markham, Ontario
  - Site 11-105, Québec, Quebec
  - Site 11-101, Saint-Jérôme, Quebec
- Georgia (6):
  - Site 59-106, Batumi
  - Site 59-102, Tbilisi
  - Site 59-104, Tbilisi
  - Site 59-103, Tbilisi
  - Site 59-105, Tbilisi
  - Site 59-107, Tbilisi
- Poland (6):
  - Site 30-107, Krakow, Malopolska
  - Site 30-104, Rzeszów, Podkarpackie Voivodeship
  - Site 30-108, Katowice, Silesian Voivodeship
  - Site 30-103, Ossy, Silesian Voivodeship
  - Site 30-109, Lodz
  - Site 30-106, Olsztyn

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who had a clinically confirmed diagnosis of hidradenitis suppurativa (HS) with a disease duration of at least 6 months before Day 1, were enrolled in the study. Randomization was stratified based on Hurley Stage at Baseline (Stage II or III).
Pre-assignment Details: 227 participants were screened for eligibility and 149 participants were randomized into the study.
Groups:
- Imsidolimab 400/200 mg: Placebo-controlled period: Participants received a starting dose of 400 milligrams (mg) of imsidolimab on Day 1 followed by 200 mg imsidolimab every 4 weeks (Days 29, 57 and 85) by subcutaneous (SC) injection. The placebo-controlled period ended at Day 113 (Week 16).
  Extension period: Participants received imsidolimab at the same dose as placebo-controlled period, SC every 4 weeks (Days 113, 141, 169, and 197).
  After discontinuation from treatment, participants remained in the study for safety follow-up period of 8 weeks.
- Imsidolimab 200/100 mg: Placebo-controlled period: Participants received a starting dose of 200 mg of imsidolimab on Day 1 followed by 100 mg imsidolimab every 4 weeks (Days 29, 57 and 85) by SC injection. The placebo-controlled period ended at Day 113 (Week 16).
  Extension period: Participants received imsidolimab at the same dose as placebo-controlled period, SC every 4 weeks (Days 113, 141, 169, and 197).
  After discontinuation from treatment, participants remained in the study for safety follow-up period of 8 weeks.
Period: Placebo-controlled Period (16 Weeks)
Arm/Group | Imsidolimab 400/200 mg | Imsidolimab 200/100 mg | Placebo
Started | 50 | 50 | 49
Completed | 41 | 42 | 43
Not Completed | 9 | 8 | 6
Not completed — Withdrawal by Subject | 6 | 5 | 4
Not completed — Lost to Follow-up | 3 | 1 | 0
Not completed — Pregnancy | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Use of Any Prohibited Medication or Treatment | 0 | 1 | 0
Period: Extension Period (16 Weeks)
Arm/Group | Imsidolimab 400/200 mg | Imsidolimab 200/100 mg | Placebo
Started | 41 | 42 | 43
Completed | 28 | 32 | 35
Not Completed | 13 | 10 | 8
Not completed — Withdrawal by Subject | 9 | 5 | 1
Not completed — Lost to Follow-up | 2 | 5 | 1
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Pregnancy | 0 | 0 | 2
Not completed — Use of Any Prohibited Medication or Treatment | 1 | 0 | 0
Not completed — Stopped participation by Sponsor | 0 | 0 | 2
Not completed — Other than specified | 0 | 0 | 1
Period: Follow-up Period (8 Weeks)
Arm/Group | Imsidolimab 400/200 mg | Imsidolimab 200/100 mg | Placebo
Started | 28 | 32 | 35
Completed | 13 | 18 | 13
Not Completed | 15 | 14 | 22
Not completed — Withdrawal by Subject | 3 | 2 | 3
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Stopped participation by Sponsor | 12 | 12 | 17

BASELINE CHARACTERISTICS:
Population: Intent to Treat (IIT) Analysis Set included all the randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Imsidolimab 400/200 mg | Imsidolimab 200/100 mg | Placebo | Total
Number analyzed (Participants) | 50 | 50 | 49 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.2 (11.35) | 36.0 (12.20) | 36.8 (11.56) | 35.7 (11.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 37 | 28 | 96
  Male | 19 | 13 | 21 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 9 | 6 | 22
  Not Hispanic or Latino | 43 | 41 | 43 | 127
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 1 | 3 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 12 | 7 | 10 | 29
  White | 36 | 37 | 37 | 110
  More than one race | 1 | 2 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 5 | 4 | 6 | 15
  United States | 29 | 29 | 30 | 88
  Poland | 11 | 15 | 13 | 39
  Georgia | 5 | 2 | 0 | 7
Abscess and Inflammatory Nodule (AN) Count [Mean (Standard Deviation); unit: count of abscess and inflammatory nodule] — The AN count was defined as the sum of the number of abscesses and inflammatory nodules from all locations.
  count of abscess and inflammatory nodule | 14.0 (9.87) | 11.9 (9.79) | 12.1 (8.31) | 12.7 (9.34)
Worst Pain Numeric Rating Scale (NRS) Score [Mean (Standard Deviation); unit: units on a scale] — Participants were asked to assign a numerical score representing the HS worst pain intensity over the last 24 hours on a scale from 0 (no symptoms) to 10 (worst imaginable symptoms). Population: ITT Analysis Set with available data was analyzed; change and percent change in worst HS pain NRS and change and percent change in average HS pain NRS are 2 different CRF questions, and so the number of responses can (and do) differ between the questions at baseline.
  units on a scale
    number analyzed (Participants) | 49 | 49 | 49 | 147
    (all) | 5.3 (2.54) | 5.4 (2.81) | 5.6 (2.79) | 5.4 (2.70)
Average pain NRS Score [Mean (Standard Deviation); unit: units on a scale] — Participants were asked to assign a numerical score representing the average intensity over the last 7 days of their HS pain symptoms on a scale from 0 (no symptoms) to 10 (worst imaginable symptoms). Population: ITT Analysis Set with available data was analyzed; change and percent change in worst HS pain NRS and change and percent change in average HS pain NRS are 2 different CRF questions, and so the number of responses can (and do) differ between the questions at baseline.
  units on a scale
    number analyzed (Participants) | 49 | 50 | 49 | 148
    (all) | 5.7 (2.61) | 6.0 (2.71) | 5.7 (2.60) | 5.8 (2.63)
Hurley Stage [Count of Participants; unit: Participants] — The Hurley system describes 3 clinical stages of HS (Stage I, II, and II). Stage I - abscess formation, single or multiple, without sinus tracts and cicatrization; Stage II - single or multiple, widely separated, recurrent abscesses with tract formation and cicatrization; Stage III - diffuse or near-diffuse involvement, or multiple interconnected tracts and abscesses across the entire area. Number of participants with Hurley Stage II and III was planned to be reported.
  Participants
    Hurley Stage Il | 36 | 38 | 37 | 111
    Hurley Stage IIl | 14 | 12 | 12 | 38

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in AN Count at Week 16: Placebo-Controlled Period
Description: The AN count was defined as the sum of the number of abscesses and inflammatory nodules from all locations.
Time Frame: Baseline, Week 16
Population: ITT Analysis Set with available data was analyzed.
Measure: Mean (Standard Deviation); unit: count of abscess and inflammatory nodule
Groups:
- Placebo-Controlled Period: Imsidolimab 400/200 mg: Participants received a starting dose of 400 mg of imsidolimab on Day 1 followed by 200 mg imsidolimab every 4 weeks (Days 29, 57 and 85) by SC injection.
- Placebo-Controlled Period: Imsidolimab 200/100 mg: Participants received a starting dose of 200 mg of imsidolimab on Day 1 followed by 100 mg imsidolimab every 4 weeks (Days 29, 57 and 85) by SC injection.
- Placebo-Controlled Period: Placebo: Participants received imsidolimab matching placebo on Day 1 and thereafter, every 4 weeks (Days 29, 57 and 85) by SC injection.
Arm/Group | Placebo-Controlled Period: Imsidolimab 400/200 mg | Placebo-Controlled Period: Imsidolimab 200/100 mg | Placebo-Controlled Period: Placebo
Number analyzed (Participants) | 39 | 41 | 42
count of abscess and inflammatory nodule | -5.9 (6.05) | -4.1 (4.63) | -5.6 (7.40)
Statistical Analysis 1: Comparison: Placebo-Controlled Period: Imsidolimab 400/200 mg vs Placebo-Controlled Period: Placebo; Test type: Superiority; p = 0.7841, Linear repeated measures model (LRMM) — LS Mean, Standard error, 90% CI, p-value based on LRMM which included: treatment, visit, treatment by visit interaction, and Hurley Stage at baseline (II vs. III) as categorical covariates; baseline AN count as continuous covariate; Least Square (LS) Mean Difference = -0.3, 90% CI 2-sided [-2.42 to 1.73], Standard Error of Mean 1.25
Statistical Analysis 2: Comparison: Placebo-Controlled Period: Imsidolimab 200/100 mg vs Placebo-Controlled Period: Placebo; Test type: Superiority; p = 0.2885, LRMM — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = 1.3, 90% CI 2-sided [-0.74 to 3.40], Standard Error of Mean 1.25

2. Secondary Outcome: Percent Change From Baseline in AN Count at Week 16: Placebo-Controlled Period
Description: The AN count was defined as the sum of the number of abscesses and inflammatory nodules from all locations.
Time Frame: Baseline, Week 16
Population: ITT Analysis Set with available data was analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo-Controlled Period: Imsidolimab 400/200 mg | Placebo-Controlled Period: Imsidolimab 200/100 mg | Placebo-Controlled Period: Placebo
Number analyzed (Participants) | 39 | 41 | 42
percent change | -44.7 (39.23) | -36.7 (36.59) | -41.2 (43.69)
Statistical Analysis 1: Comparison: Placebo-Controlled Period: Imsidolimab 400/200 mg vs Placebo-Controlled Period: Placebo; Test type: Superiority; p = 0.5939, LRMM — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -4.8, 90% CI 2-sided [-19.66 to 10.07], Standard Error of Mean 8.97
Statistical Analysis 2: Comparison: Placebo-Controlled Period: Imsidolimab 200/100 mg vs Placebo-Controlled Period: Placebo; Test type: Superiority; p = 0.7002, LRMM — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = 3.5, 90% CI 2-sided [-11.38 to 18.29], Standard Error of Mean 8.95

3. Secondary Outcome: Number of Participants Achieving Hidradenitis Suppurativa Clinical Response 50 (HiSCR50): Placebo-Controlled Period
Description: The number of participants with at least a 50% decrease from Baseline AN count, and no increase in abscesses or draining fistulas in comparison to baseline (HiSCR50) at Week 16 was calculated for each treatment group as follows:
  A responder HiSCR50 was defined as a participant with
  1. at least a 50% decrease in AN count from Baseline, and
  2. no increase in abscess count relative to Baseline, and
  3. no increase in draining fistula count relative to Baseline
Time Frame: Week 16
Population: ITT Analysis Set with available data was analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Controlled Period: Imsidolimab 400/200 mg | Placebo-Controlled Period: Imsidolimab 200/100 mg | Placebo-Controlled Period: Placebo
Number analyzed (Participants) | 39 | 41 | 42
Participants | 16 | 16 | 15
Statistical Analysis 1: Comparison: Placebo-Controlled Period: Imsidolimab 400/200 mg vs Placebo-Controlled Period: Placebo; Test type: Superiority; Risk Difference (RD) = 5.3, 90% CI 2-sided [-13.3 to 23.4] — Estimate parameter and 90% CI was based on Unadjusted Risk Difference and exact unconditional confidence intervals (CI)
Statistical Analysis 2: Comparison: Placebo-Controlled Period: Imsidolimab 200/100 mg vs Placebo-Controlled Period: Placebo; Test type: Superiority; Risk Difference (RD) = 3.3, 90% CI 2-sided [-14.6 to 21.0] — Estimate parameter and 90% C was based on Unadjusted Risk Difference and exact unconditional CIs

4. Secondary Outcome: Change From Baseline in Worst HS Pain NRS Score at Week 16: Placebo-Controlled Period
Description: Participants were asked to assign a numerical score representing the HS worst pain intensity over the last 24 hours on a scale from 0 (no symptoms) to 10 (worst imaginable symptoms).
Time Frame: Baseline, Week 16
Population: ITT Analysis Set with available data was analyzed; change and percent change in worst HS pain NRS and change and percent change in average HS pain NRS are 2 different CRF questions, and so the number of responses can (and do) differ between the questions at baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo-Controlled Period: Imsidolimab 400/200 mg | Placebo-Controlled Period: Imsidolimab 200/100 mg | Placebo-Controlled Period: Placebo
Number analyzed (Participants) | 39 | 40 | 42
units on a scale | -0.3 (2.89) | -0.7 (2.37) | -0.4 (3.22)
Statistical Analysis 1: Comparison: Placebo-Controlled Period: Imsidolimab 400/200 mg vs Placebo-Controlled Period: Placebo; Test type: Superiority; p = 0.7282, LRMM — LS Mean, Standard error, 90% CI, p-value based on LRMM which included: treatment, visit, treatment by visit interaction, and Hurley Stage at baseline (II vs. III) as categorical covariates and baseline worst HS Pain NRS as a continuous covariate; LS Mean Difference = -0.2, 90% CI 2-sided [-1.08 to 0.70], Standard Error of Mean 0.54
Statistical Analysis 2: Comparison: Placebo-Controlled Period: Imsidolimab 200/100 mg vs Placebo-Controlled Period: Placebo; Test type: Superiority; p = 0.5019, LRMM — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = -0.4, 90% CI 2-sided [-1.25 to 0.53], Standard Error of Mean 0.54

5. Secondary Outcome: Change From Baseline in Average HS Pain NRS Score at Week 16: Placebo-Controlled Period
Description: Participants were asked to assign a numerical score representing the average intensity over the last 7 days of their HS pain symptoms on a scale from 0 (no symptoms) to 10 (worst imaginable symptoms).
Time Frame: Baseline, Week 16
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo-Controlled Period: Imsidolimab 400/200 mg | Placebo-Controlled Period: Imsidolimab 200/100 mg | Placebo-Controlled Period: Placebo
Number analyzed (Participants) | 39 | 41 | 42
units on a scale | -0.5 (2.29) | -1.0 (2.48) | -0.5 (2.74)
Statistical Analysis 1: Comparison: Placebo-Controlled Period: Imsidolimab 400/200 mg vs Placebo-Controlled Period: Placebo; Test type: Superiority; p = 0.7698, LRMM — LS Mean, Standard error, 90% CI, p-value based on LRMM which included: treatment, visit, treatment by visit interaction, and Hurley Stage at baseline (II vs. III) as categorical covariates and baseline average HS Pain NRS as a continuous covariate; LS Mean Difference = -0.1, 90% CI 2-sided [-0.96 to 0.67], Standard Error of Mean 0.49
Statistical Analysis 2: Comparison: Placebo-Controlled Period: Imsidolimab 200/100 mg vs Placebo-Controlled Period: Placebo; Test type: Superiority; p = 0.7468, LRMM — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -0.2, 90% CI 2-sided [-0.97 to 0.65], Standard Error of Mean 0.49

6. Secondary Outcome: Percent Change From Baseline in Worst HS Pain NRS Score at Week 16: Placebo-Controlled Period
Description: Participants were asked to assign a numerical score representing the HS worst pain intensity over the last 24 hours on a scale from 0 (no symptoms) to 10 (worst imaginable symptoms). Only participants that had Baseline score of >0 could be included in the analysis of Percent Change from Baseline.
Time Frame: Baseline, Week 16
Population: ITT Analysis Set with available data was analyzed; change and percent change in worst HS pain NRS and change and percent change in average HS pain NRS are 2 different CRF questions, and so the number of responses can (and do) differ between the questions at baseline. "Overall number of participants analyzed" included only those participants with Baseline score of >0.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo-Controlled Period: Imsidolimab 400/200 mg | Placebo-Controlled Period: Imsidolimab 200/100 mg | Placebo-Controlled Period: Placebo
Number analyzed (Participants) | 37 | 38 | 40
percent change | 7.6 (81.81) | 10.2 (146.92) | 30.3 (136.89)
Statistical Analysis 1: Comparison: Placebo-Controlled Period: Imsidolimab 400/200 mg vs Placebo-Controlled Period: Placebo; Test type: Superiority; p = 0.2750, LRMM — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = -25.7, 90% CI 2-sided [-64.57 to 13.14], Standard Error of Mean 23.46
Statistical Analysis 2: Comparison: Placebo-Controlled Period: Imsidolimab 200/100 mg vs Placebo-Controlled Period: Placebo; Test type: Superiority; p = 0.3757, LRMM — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = -21.2, 90% CI 2-sided [-60.60 to 18.28], Standard Error of Mean 23.81

7. Secondary Outcome: Percent Change From Baseline in Average HS Pain NRS Score at Week 16: Placebo-Controlled Period
Description: Participants were asked to assign a numerical score representing the average intensity over the last 7 days of their HS pain symptoms on a scale from 0 (no symptoms) to 10 (worst imaginable symptoms). Only participants that had Baseline score of >0 could be included in the analysis of Percent Change from Baseline.
Time Frame: Baseline, Week 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo-Controlled Period: Imsidolimab 400/200 mg | Placebo-Controlled Period: Imsidolimab 200/100 mg | Placebo-Controlled Period: Placebo
Number analyzed (Participants) | 37 | 39 | 41
percent change | -1.3 (58.54) | -18.3 (37.76) | 4.5 (77.25)
Statistical Analysis 1: Comparison: Placebo-Controlled Period: Imsidolimab 400/200 mg vs Placebo-Controlled Period: Placebo; Test type: Superiority; p = 0.6146, LRMM — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -6.6, 90% CI 2-sided [-28.22 to 15.05], Standard Error of Mean 13.04
Statistical Analysis 2: Comparison: Placebo-Controlled Period: Imsidolimab 200/100 mg vs Placebo-Controlled Period: Placebo; Test type: Superiority; p = 0.4951, LRMM — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -8.9, 90% CI 2-sided [-30.35 to 12.62], Standard Error of Mean 12.95

8. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs): Placebo-Controlled Period
Description: An adverse event (AE) was any untoward medical occurrence in a participant temporally associated with the use of a study treatment, whether or not considered related to the study treatment. An AE was considered treatment-emergent if the date of onset was during or after first dose of study treatment during placebo-controlled period, or if the AE present at baseline worsened in either intensity or frequency after first dose of study treatment.
Time Frame: From first dose (placebo-controlled period) up to Week 16
Population: Safety analysis set included all randomized participants who received at least 1 dose of imsidolimab or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Controlled Period: Imsidolimab 400/200 mg | Placebo-Controlled Period: Imsidolimab 200/100 mg | Placebo-Controlled Period: Placebo
Number analyzed (Participants) | 50 | 50 | 49
Participants | 19 | 14 | 18

9. Secondary Outcome: Number of Participants With TEAEs: Extension and Follow-up Period
Description: An AE was any untoward medical occurrence in a participant temporally associated with the use of a study treatment, whether or not considered related to the study treatment. An AE was considered treatment-emergent if the date of onset was during or after first dose of study treatment in extension period, or if the AE present at baseline worsened in either intensity or frequency after first dose of study treatment.
Time Frame: From first dose (extension period) up to Week 40
Population: Extension Analysis Set included subset of the safety analysis set who received at least 1 dose of imsidolimab in the extension period.
Measure: Count of Participants; unit: Participants
Groups:
- Extension Period: Imsidolimab 400/200 mg: Participants received a dose of 400 mg of imsidolimab on Day 113, followed by a 200-mg dose on Days 141, 169, and 197 by SC injection.
- Extension Period: Imsidolimab 200/100 mg: Participants received a dose of 200 mg of imsidolimab on Day 113, followed by a 100-mg dose on Days 141, 169, and 197 by SC injection.
- Extension Period: Placebo to Imsidolimab 400/200 mg: Participants who received placebo in placebo-controlled period, received 400 mg of imsidolimab on Day 113, followed by a dose of 200 mg on Days 141, 169, and 197 by SC injection in extension period.
- Extension Period: Placebo to Imsidolimab 200/100 mg: Participants who received placebo in placebo-controlled period, received 200 mg of imsidolimab on Day 113, followed by a dose of 100 mg on Days 141, 169, and 197 by SC injection in extension period.
Arm/Group | Extension Period: Imsidolimab 400/200 mg | Extension Period: Imsidolimab 200/100 mg | Extension Period: Placebo to Imsidolimab 400/200 mg | Extension Period: Placebo to Imsidolimab 200/100 mg
Number analyzed (Participants) | 40 | 42 | 19 | 21
Participants | 15 | 18 | 9 | 10

ADVERSE EVENTS:
Time Frame: From first dose up to Week 40
Description: Placebo-Controlled Period: Safety Analysis Set
  Extension Period: Extension Analysis Set
Groups:
- Extension Period: Imsidolimab 400/200 mg: Participants received a dose of 400 mg of imsidolimab on Day 113, followed by a dose of 200 mg on Days 141, 169, and 197 by SC injection.
- Extension Period: Imsidolimab 200/100 mg: Participants received a dose of 200 mg of imsidolimab on Day 113, followed by a dose of 100 mg on Days 141, 169, and 197 by SC injection.
Arm/Group | Placebo-Controlled Period: Imsidolimab 400/200 mg | Placebo-Controlled Period: Imsidolimab 200/100 mg | Placebo-Controlled Period: Placebo | Extension Period: Imsidolimab 400/200 mg | Extension Period: Imsidolimab 200/100 mg | Extension Period: Placebo to Imsidolimab 400/200 mg | Extension Period: Placebo to Imsidolimab 200/100 mg
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50 | 0/49 | 0/40 | 0/42 | 0/19 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/50 | 2/50 | 3/49 | 0/40 | 1/42 | 0/19 | 0/21
Other Adverse Events (participants affected / at risk) | 5/50 | 6/50 | 9/49 | 9/40 | 10/42 | 9/19 | 5/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo-Controlled Period: Imsidolimab 400/200 mg (N=50) | Placebo-Controlled Period: Imsidolimab 200/100 mg (N=50) | Placebo-Controlled Period: Placebo (N=49) | Extension Period: Imsidolimab 400/200 mg (N=40) | Extension Period: Imsidolimab 200/100 mg (N=42) | Extension Period: Placebo to Imsidolimab 400/200 mg (N=19) | Extension Period: Placebo to Imsidolimab 200/100 mg (N=21)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo-Controlled Period: Imsidolimab 400/200 mg (N=50) | Placebo-Controlled Period: Imsidolimab 200/100 mg (N=50) | Placebo-Controlled Period: Placebo (N=49) | Extension Period: Imsidolimab 400/200 mg (N=40) | Extension Period: Imsidolimab 200/100 mg (N=42) | Extension Period: Placebo to Imsidolimab 400/200 mg (N=19) | Extension Period: Placebo to Imsidolimab 200/100 mg (N=21)
COVID-19 (Infections and infestations) | 4 (4) | 3 (3) | 3 (3) | 2 (2) | 3 (3) | 0 (0) | 3 (3)
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 4 (6) | 3 (4) | 2 (2) | 1 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia areata (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-09-24): https://cdn.clinicaltrials.gov/large-docs/30/NCT04856930/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-16): https://cdn.clinicaltrials.gov/large-docs/30/NCT04856930/SAP_001.pdf